CLINICAL TRIAL: NCT01717742
Title: Intrapleural DNase and Tissue Plasminogen Activator in Pediatric Empyema (DTPA Trial)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Children's Hospital of Eastern Ontario (Other); St. Justine's Hospital (Other); Unity Health Toronto (Other); The Physicians' Services Incorporated Foundation (Other); McMaster Children's Hospital (Other); British Columbia Children's Hospital (Other)
Responsible Party: Principal Investigator, Eyal Cohen, Staff Physician, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1000033767
Record Dates: First submitted 2012-10-25; First posted 2012-10-30 (Estimated); Results first posted 2020-04-03 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Pleural Empyema
Keywords: Randomized controlled trial; Pleural Empyema; tPA; DNase
MeSH Terms: conditions — Empyema, Pleural | interventions — Tissue Plasminogen Activator; Deoxyribonucleases; dornase alfa; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- tPA and placebo (Active Comparator)
  Interventions: Drug: TPA (Tissue Plasminogen Activator); Other: Placebo
- tPA and DNase (Experimental)
  Interventions: Drug: TPA (Tissue Plasminogen Activator); Drug: DNase

INTERVENTIONS:
Drug: TPA (Tissue Plasminogen Activator) — Intrapleural administration of tPA 4 mg in 10 ml (≤10 kg) or 20 ml (>10 kg) normal saline once daily for 3 days
  Other Names: Cathflo (alteplase, recombinant)
Drug: DNase — Intrapleural administration of DNase 5 mg diluted to 10 ml (≤10 kg) or 20 ml (>10 kg) normal saline once daily for 3 days
  Other Names: Pulmozyme (Dornase alfa)
  Arms: tPA and DNase
Other: Placebo — Intrapleural administration of normal saline 10 ml (≤10 kg) or 20 ml (>10 kg)
  Other Names: Normal saline
  Arms: tPA and placebo

SUMMARY:
Bacterial pneumonia can be complicated by the development of excess fluid and pus (pleural empyema) around the lungs in children. The incidence of pleural empyema in children has increased significantly in the last 10 years.

Short term morbidity for this condition is substantial, but unlike in adults, the long term outcome of this condition for children in developed countries is favourable. Inserting a chest drain and then adding a medicine (tissue plasminogen activator - tPA) to break down organized pus has been shown to be an effective therapy for reducing the duration of illness. However, this treatment is still suboptimal and prolonged hospitalization is common. Recent data from adults suggests that adding an additional medicine (DNase) to decrease the viscosity (thickness) of the fluid improves drainage and leads to better patient outcomes; however, there are no published studies on children.

This is a multi-centre randomized controlled trial comparing the time to discharge from hospital after chest drain insertion in previously well children who present with pleural empyema, treated with intrapleural DNase and tissue plasminogen activator (tPA) by chest drain for three doses over 48 hours compared with three doses over 48 hours of tPA alone. Other outcomes related to effectiveness, safety and cost will be assessed as well.

ELIGIBILITY:
Inclusion Criteria:

1. age 6 months to 18 years
2. hospitalized with diagnosis of pleural empyema requiring chest tube drainage with fibrinolytics as judged by the attending physician with the following criteria:

   1. pneumonia with pleural effusion as documented on ultrasound of the chest; AND
   2. need for further intervention in addition to antibiotics based on clinical criteria [persistent fever despite on antibiotics for at least 48 hours OR significant respiratory distress tachypnea, hypoxia) as a result of the pleural fluid collection]

Exclusion Criteria:

1. empyema as a result of tuberculosis, fungus or non-infectious causes (e.g. malignancy)
2. known coagulation impairment
3. suspected or proven allergy to tPA or DNase
4. chronic lung disease or other chronic illnesses (e.g. immunodeficiency or neurologic impairment)
5. child has already undergone a drainage procedure (e.g. chest drain or VATS).
6. recent administration of an investigational drug (within previous 30 days)
7. pregnancy
8. breastfeeding

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 97 (Actual)
Dates: Start 2012-12; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eyal Cohen, MD, MSc, Principal Investigator — The Hospital for Sick Children
Locations (6):
- Canada (6):
  - Alberta Children's Hospital, Calgary, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - McMaster Children's Hospital, Hamilton, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - The Hospital for Sick Children(SickKids), Toronto, Ontario
  - CHU Sainte Justine, Montreal, Quebec

REFERENCES:
- [Result] Livingston MH, Mahant S, Connolly B, MacLusky I, Laberge S, Giglia L, Yang C, Roberts A, Shawyer A, Brindle M, Parsons S, Stoian C, Walton JM, Thorpe KE, Chen Y, Zuo F, Mamdani M, Chan C, Loong D, Isaranuwatchai W, Ratjen F, Cohen E. Effectiveness of Intrapleural Tissue Plasminogen Activator and Dornase Alfa vs Tissue Plasminogen Activator Alone in Children with Pleural Empyema: A Randomized Clinical Trial. JAMA Pediatr. 2020 Apr 1;174(4):332-340. doi: 10.1001/jamapediatrics.2019.5863. PMID 32011642
- [Derived] Livingston MH, Mahant S, Ratjen F, Connolly BL, Thorpe K, Mamdani M, Maclusky I, Laberge S, Giglia L, Walton JM, Yang CL, Roberts A, Shawyer AC, Brindle M, Parsons SJ, Stoian CA, Cohen E. Intrapleural Dornase and Tissue Plasminogen Activator in pediatric empyema (DTPA): a study protocol for a randomized controlled trial. Trials. 2017 Jun 24;18(1):293. doi: 10.1186/s13063-017-2026-0. PMID 28646887

RESULTS

PARTICIPANT FLOW:
Groups:
- tPA (Tissue Plasminogen Activator) and Placebo: tPA: Intrapleural administration of tPA 4 mg in 10 ml (≤10 kg) or 20 ml (>10 kg) normal saline once daily for 3 days
  Placebo: Intrapleural administration of normal saline 10 ml (≤10 kg) or 20 ml (>10 kg)
- tPA (Tissue Plasminogen Activator) and DNase: tPA: Intrapleural administration of tPA 4 mg in 10 ml (≤10 kg) or 20 ml (>10 kg) normal saline once daily for 3 days
  DNase: Intrapleural administration of DNase 5 mg diluted to 10 ml (≤10 kg) or 20 ml (>10 kg) normal saline once daily for 3 days
Period: Overall Study
Arm/Group | tPA (Tissue Plasminogen Activator) and Placebo | tPA (Tissue Plasminogen Activator) and DNase
Started | 48 | 49
Completed | 43 | 47
Not Completed | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Intervention (tPA & DNase): Intrapleural tPA, 4 mg, followed by DNase (Roche), 5 mg
- Placebo (tPA & Placebo): Intrapleural tPA (Roche), 4 mg, followed by 5 mL of normal saline
- Total: Total of all reporting groups
Arm/Group | Intervention (tPA & DNase) | Placebo (tPA & Placebo) | Total
Number analyzed (Participants) | 49 | 48 | 97
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 49 | 48 | 97
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Months] | 58.4 (43.3) | 64.1 (44.2) | 61.3 (45.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 21 | 45
  Male | 25 | 27 | 52
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/ethnicity: First nations | 0 | 2 | 2
  Race/ethnicity: African | 2 | 0 | 2
  Race/ethnicity: Asian/Pacific Islander | 14 | 13 | 27
  Race/ethnicity: White | 26 | 26 | 52
  Race/ethnicity: Hispanic | 1 | 0 | 1
  Race/ethnicity: Middle Eastern | 0 | 1 | 1
  Race/ethnicity: South Asian | 0 | 1 | 1
  Race/ethnicity: Prefer not to answer | 5 | 4 | 9
  Race/ethnicity: Missing | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 49 | 48 | 97

OUTCOME MEASURES:

1. Primary Outcome: Time to Hospital Discharge
Description: Time from insertion of the chest drain to discharge from hospital.
Time Frame: up to 4 months
Measure: Mean (Standard Deviation); unit: days
Groups:
- Intervention: Intervention group received intrapleural tPA, 4 mg, followed by DNase (Roche), 5 mg
- Control: Control group received intrapleural tPA (Roche), 4 mg, followed by 5 mL of normal saline
Arm/Group | Intervention | Control
Number analyzed (Participants) | 49 | 48
days | 9.0 (4.9) | 9.1 (5.3)

2. Secondary Outcome: Time to Meeting Discharge Criteria
Description: Time from insertion of the chest drain to meeting discharge criteria.
  Discharge criteria:
  * Chest tube removed
  * No fever [temperature less than 38°C]
  * Normal respiratory rate forage
  * No hypoxia
  * Drinking fluids wel
Time Frame: up to 4 months
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Intervention | Control
Number analyzed (Participants) | 49 | 48
days | 8.2 (4.5) | 8.5 (5.4)

3. Secondary Outcome: Time to Drain Removal
Description: Time from drain insertion to drain removal.
Time Frame: up to 4 months
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Intervention | Control
Number analyzed (Participants) | 49 | 48
days | 6.9 (4.3) | 6.9 (5.3)

4. Secondary Outcome: Duration of Fever After Intervention
Description: Duration of fever (defined as temperature >38 degrees celsius taken by any method) from insertion of the chest drain until resolution.
Time Frame: up to 4 months
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Intervention | Control
Number analyzed (Participants) | 49 | 48
days | 2.8 (3.4) | 3.3 (3.4)

5. Secondary Outcome: Number of Participants With Need for Ventilatory Support or Non-invasive Ventilation Following the Intervention
Description: Number of Participants with need for any kind of ventilatory support or any kind of non-invasive ventilation right after the intervention.
Time Frame: up to 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 49 | 48
Participants | 9 | 8

6. Secondary Outcome: Number of Participants With Serious Bleeding
Description: Number of Participants who had intrapleural bleeding resulting in a drop in hemoglobin of greater than 20 g/L or needing a transfusion.
Time Frame: up to 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 49 | 48
Participants | 2 | 4

7. Secondary Outcome: Number of Participants With Further Interventions
Description: Number of participants who needed further intervention such as placement of another chest drain (by any technique) or surgical intervention such as thoracotomy and decortication, video-assisted thorascopic surgery, or pneumonectomy.
Time Frame: up to 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 49 | 48
Participants | 4 | 2

8. Secondary Outcome: Number of Participants With Hospital Readmission
Description: Number of Participants who had any hospital readmission after discharge from hospital for initial treatment for pleural empyema within three months related to pleural empyema or its treatment.
Time Frame: 3 months post-discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 49 | 48
Participants | 2 | 0

9. Secondary Outcome: Cost of the Hospitalization
Description: An economic evaluation will compare the relative costs of DNase-tPA with tPA alone in previously well children who present with pleural empyema, using patient-level data from the trial.
Time Frame: up to 4 months
Measure: Mean (Standard Deviation); unit: 2018 US $
Arm/Group | Intervention | Control
Number analyzed (Participants) | 49 | 48
2018 US $ | 11329 (7139) | 10760 (5071)

10. Secondary Outcome: Mortality
Description: Mortality from any cause during the hospitalization for empyema.
Time Frame: up to 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 49 | 48
Participants | 0 | 0

11. Other Pre Specified Outcome: Chest Radiography
Description: The radiograph closest to the time of drain removal will be reviewed by a blinded study radiologist to determine the percentage of hemithorax occupied using a 5 point ordinal scale utilized in previous studies ranging from no fluid present to fluid occupying >75% of the most affected hemithorax.
Time Frame: 7 days after drain removal
Population: Degree of opacification on chest radiography prior to chest tube removal
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 49 | 48
Participants
  <=25% | 33 | 25
  26-50% | 10 | 11
  51-75% | 1 | 4
  >75% | 2 | 1
  Missing | 3 | 7

ADVERSE EVENTS:
Time Frame: Over the course of the patient's hospitalization
Description: All serious unexpected adverse events were reported to the REB. All serious adverse drug reactions to the study medication were reported to Health Canada within 15 calendar days or for death or life-threatening events, within 7 calendar days. In the latter case, a follow-up report was filed within 8 calendar days. Adverse reactions will be managed according to the standard clinical management practices. All adverse events and adverse reactions were reported to the PI within 24 hours.
Groups:
- Intervention: Intervention group received ) intrapleural tPA, 4 mg, followed by DNase (Roche), 5 mg
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/48
Serious Adverse Events (participants affected / at risk) | 6/49 | 8/48
Other Adverse Events (participants affected / at risk) | 8/49 | 13/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=49) | Control (N=48)
TENSION PYOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Serious bleeding (Blood and lymphatic system disorders) | 2 (2) | 4 (4)
Bronchopleural fistula (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Hemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Low hemoglobin levels (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Septic shock (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=49) | Control (N=48)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2)
Edema (General disorders) | 0 (0) | 2 (2)
Transient chest pain (Cardiac disorders) | 1 (1) | 0 (0)
Herpes simplex virus infection (Immune system disorders) | 1 (1) | 0 (0)
Mild bleeding (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Kinked chest tube (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Low albumin (Endocrine disorders) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Other bacterial infection (Immune system disorders) | 1 (1) | 0 (0)
Chest tube removed accidentally (General disorders) | 0 (0) | 1 (1)
Elevated potassium (Endocrine disorders) | 0 (0) | 1 (1)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Urinary infection (Renal and urinary disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-06-29): https://cdn.clinicaltrials.gov/large-docs/42/NCT01717742/Prot_SAP_000.pdf
  • Informed Consent Form (2017-10-12): https://cdn.clinicaltrials.gov/large-docs/42/NCT01717742/ICF_001.pdf